CLINICAL TRIAL: NCT00932672
Title: Randomized Controlled Clinical Trial of Carbohydrate Restriction Among Men Initiating Androgen Deprivation Therapy For Prostate Cancer
Brief Title: Atkins Diet and Prostate Cancer Clinical Trial
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow recruitment, lack of funding and PI transferred
Sponsor: Duke University (Other)
Collaborators: VA Greater Los Angeles Healthcare System (U.S. Federal Agency); Durham VA Medical Center (U.S. Federal Agency); University of California, Los Angeles (Other); Carolina Urologic Research Center (Other); First Urology (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00010519
Record Dates: First submitted 2009-07-02; First posted 2009-07-03 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-12

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Atkins
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Diet, High-Protein Low-Carbohydrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atkins group (Experimental): Men assigned to the Atkins diet will be asked to restrict carbohydrate intake to <20 grams/day. We will use an established clinical program directed by Dr. Eric Westman which implements this diet using a trained clinical nutritionist. No other dietary restrictions will be placed on the subjects. They will measure their urinary ketones at home weekly using urinary ketone strips. Subjects will meet with the nutritionist monthly during the 6 months of the study. Subjects in the Atkins arm will also be asked to walk at a brisk pace for 30 minutes a day, 5 days a week and will be provided a pedometer to measure the number of steps taken per day.
  Interventions: Behavioral: Atkins Diet
- Control group (No Intervention): Subjects assigned to the control group will be asked to make no changes in their dietary habits. At the completion of the study subjects will meet with the nutritionist and receive standard nutrition AHA recommendations.

INTERVENTIONS:
Behavioral: Atkins Diet — Patients are given an outline of the Atkins diet and are asked to follow it for 6 months
  Other Names: Atkins group; Cases
  Arms: Atkins group

SUMMARY:
This study will test the hypothesis that a low-carbohydrate Atkins diet will prevent or at least minimize the metabolic consequences of androgen deprivation therapy (ADT).

DETAILED DESCRIPTION:
Androgen deprivation therapy (ADT) is the standard treatment for advanced prostate cancer. While a very effective anti-cancer treatment, ADT is associated with significant toxicity including but not limited to major metabolic disturbances including impaired glucose tolerance, insulin resistance, and weight gain. We hypothesize that limiting carbohydrates within the diet will prevent or at least minimize these consequences.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma of the prostate
2. Scheduled to initiate ADT with an anticipated duration of ≥ 6 months
3. Overweight or obese (body mass index ≥ 25 kg/m2)

Exclusion Criteria:

1. Symptomatic metastatic disease
2. Myocardial infarction within 6 months
3. Treatment with medications known to affect insulin or glucose levels (i.e. insulin, oral hypoglycemics, prednisone, etc.)
4. Patient consuming a low-carbohydrate diet
5. Medical conditions or co-morbidities that preclude participation in the protocol
6. Vegetarians

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2009-06; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
The primary end-point will be differences in insulin sensitivity between the arms | 6 months

SECONDARY OUTCOMES:
Measures will include other cardiac risk factors, overall body morphometrics, body composition as assessed by dual energy x-ray absorptiometry (DXA), and cancer control (PSA levels) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Freedland, MD, Principal Investigator — Duke University
Locations (3):
- United States (3):
  - Greater Los Angeles VA Medical Center, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - Duke University Medical Center, Durham, North Carolina

REFERENCES:
- [Background] Loblaw DA, Virgo KS, Nam R, Somerfield MR, Ben-Josef E, Mendelson DS, Middleton R, Sharp SA, Smith TJ, Talcott J, Taplin M, Vogelzang NJ, Wade JL 3rd, Bennett CL, Scher HI; American Society of Clinical Oncology. Initial hormonal management of androgen-sensitive metastatic, recurrent, or progressive prostate cancer: 2006 update of an American Society of Clinical Oncology practice guideline. J Clin Oncol. 2007 Apr 20;25(12):1596-605. doi: 10.1200/JCO.2006.10.1949. Epub 2007 Apr 2. PMID 17404365
- [Background] Bolla M, Gonzalez D, Warde P, Dubois JB, Mirimanoff RO, Storme G, Bernier J, Kuten A, Sternberg C, Gil T, Collette L, Pierart M. Improved survival in patients with locally advanced prostate cancer treated with radiotherapy and goserelin. N Engl J Med. 1997 Jul 31;337(5):295-300. doi: 10.1056/NEJM199707313370502. PMID 9233866
- [Background] Smith MR, Lee H, Nathan DM. Insulin sensitivity during combined androgen blockade for prostate cancer. J Clin Endocrinol Metab. 2006 Apr;91(4):1305-8. doi: 10.1210/jc.2005-2507. Epub 2006 Jan 24. PMID 16434464
- [Background] Keating NL, O'Malley AJ, Smith MR. Diabetes and cardiovascular disease during androgen deprivation therapy for prostate cancer. J Clin Oncol. 2006 Sep 20;24(27):4448-56. doi: 10.1200/JCO.2006.06.2497. PMID 16983113
- [Background] Tsai HK, D'Amico AV, Sadetsky N, Chen MH, Carroll PR. Androgen deprivation therapy for localized prostate cancer and the risk of cardiovascular mortality. J Natl Cancer Inst. 2007 Oct 17;99(20):1516-24. doi: 10.1093/jnci/djm168. Epub 2007 Oct 9. PMID 17925537
- [Background] D'Amico AV, Chen MH, Renshaw AA, Loffredo M, Kantoff PW. Androgen suppression and radiation vs radiation alone for prostate cancer: a randomized trial. JAMA. 2008 Jan 23;299(3):289-95. doi: 10.1001/jama.299.3.289. PMID 18212313
- [Background] Saigal CS, Gore JL, Krupski TL, Hanley J, Schonlau M, Litwin MS; Urologic Diseases in America Project. Androgen deprivation therapy increases cardiovascular morbidity in men with prostate cancer. Cancer. 2007 Oct 1;110(7):1493-500. doi: 10.1002/cncr.22933. PMID 17657815
- [Background] Gardner CD, Kiazand A, Alhassan S, Kim S, Stafford RS, Balise RR, Kraemer HC, King AC. Comparison of the Atkins, Zone, Ornish, and LEARN diets for change in weight and related risk factors among overweight premenopausal women: the A TO Z Weight Loss Study: a randomized trial. JAMA. 2007 Mar 7;297(9):969-77. doi: 10.1001/jama.297.9.969. PMID 17341711
- [Background] Freedland SJ, Mavropoulos J, Wang A, Darshan M, Demark-Wahnefried W, Aronson WJ, Cohen P, Hwang D, Peterson B, Fields T, Pizzo SV, Isaacs WB. Carbohydrate restriction, prostate cancer growth, and the insulin-like growth factor axis. Prostate. 2008 Jan 1;68(1):11-9. doi: 10.1002/pros.20683. PMID 17999389
- [Background] Yancy WS Jr, Olsen MK, Guyton JR, Bakst RP, Westman EC. A low-carbohydrate, ketogenic diet versus a low-fat diet to treat obesity and hyperlipidemia: a randomized, controlled trial. Ann Intern Med. 2004 May 18;140(10):769-77. doi: 10.7326/0003-4819-140-10-200405180-00006. PMID 15148063
- [Background] Matthews DR, Hosker JP, Rudenski AS, Naylor BA, Treacher DF, Turner RC. Homeostasis model assessment: insulin resistance and beta-cell function from fasting plasma glucose and insulin concentrations in man. Diabetologia. 1985 Jul;28(7):412-9. doi: 10.1007/BF00280883. PMID 3899825
- [Background] Smith MR, Finkelstein JS, McGovern FJ, Zietman AL, Fallon MA, Schoenfeld DA, Kantoff PW. Changes in body composition during androgen deprivation therapy for prostate cancer. J Clin Endocrinol Metab. 2002 Feb;87(2):599-603. doi: 10.1210/jcem.87.2.8299. PMID 11836291
- [Background] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527
- [Background] Barry MJ, Delorenzo MA, Walker-Corkery ES, Lucas FL, Wennberg DC. The rising prevalence of androgen deprivation among older American men since the advent of prostate-specific antigen testing: a population-based cohort study. BJU Int. 2006 Nov;98(5):973-8. doi: 10.1111/j.1464-410X.2006.06416.x. Epub 2006 Jul 28. PMID 16879443
- [Derived] Freedland SJ, Howard LE, Ngo A, Ramirez-Torres A, Csizmadi I, Cheng S, Mack A, Lin PH. Low Carbohydrate Diets and Estimated Cardiovascular and Metabolic Syndrome Risk in Prostate Cancer. J Urol. 2021 Dec;206(6):1411-1419. doi: 10.1097/JU.0000000000002112. Epub 2021 Jul 14. PMID 34259565
- See also: Atkins Diet Weight Loss Program — http://www.atkins.com